CLINICAL TRIAL: NCT02041637
Title: Unknown Cause of Acute Liver Failure: Determination of Early Mortality Predictive Factors
Brief Title: Unknown Cause of Acute Liver Failure
Acronym: HASIPRO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM11030
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Liver Failure; Unknown Etiology
Keywords: liver failure; etiology; liver transplantation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate the outcome and to determine predictive factors of patients admitted in a context of acute liver failure without identified cause.

DETAILED DESCRIPTION:
Methodology: Multicentric French national cohort with prospective collection of data and constitution of biobank, in patients hospitalized in a context of acute liver failure without known cause at admission. Follow-up during 3 months for each patients. The primary objective is to determine predictive factors of early mortality. This study is an observational cohort and patients will received standard care during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Acute liver failure defined by a PT<50% or INR>1.5;
* with or without hepatic encephalopathy;
* without cause identified at admission, and non A non B hepatitis;
* age>18 year old;
* signed an informed consent.

Exclusion Criteria:

* chronic liver disease;
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute liver failure without cause identified at admission
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
mortality | At 3 months

SECONDARY OUTCOMES:
Liver transplantation rate | At 3 months
Overall survival rate | At 3 months
post-transplant mortality rate | At 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Audrey COILLY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Didier Samuel, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif, France